CLINICAL TRIAL: NCT05104073
Title: Califormula Study: Calibrated Formula Feeding to Optimize Infant Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Staff Physician Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00018788; 1R21HD104028-01 (NIH)
Record Dates: First submitted 2021-10-11; First posted 2021-11-02 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A cohort of 60 infants will be recruited and randomized 2-3 weeks after birth to an intervention arm characterized by calibrated formula feeding recommendations or a control group with ad lib feeds as per usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm is characterized by calibrated formula feeding recommendations. The intervention group parents will be given written instructions on infant hunger and satiety cues as well as copies of videos with guidance on bottle feeding and how to soothe fussy infants without feeding. N=30 meeting inclusion/exclusion criteria
  Interventions: Behavioral: Intervention
- Control (No Intervention): The control arm will have ad lib feeds as per usual care. N=30 meeting inclusion/exclusion criteria

INTERVENTIONS:
Behavioral: Intervention — Provided with educational materials, guidelines and instructions.
  Arms: Intervention

SUMMARY:
The purpose of this voluntary research study is to determine if calibrated formula feeding recommendations can promote optimal growth for the first 6 months after birth for mothers with a pre-pregnancy body mass index of 25 or more.

DETAILED DESCRIPTION:
This pilot study seeks to determine if formula feeding recommendations that are calibrated using age and weight specific caloric intake recommendations can prevent excessive infant weight gain and reduce overweight in the first 6 months after birth among infants born to mothers with overweight prior to pregnancy electing to exclusively formula feed their infants. Calibrated formula feeding refers to adjusting the recommended daily caloric formula intake to account for weight status. A cohort of 60 infants will be recruited and randomized 2-3 weeks after birth to an intervention arm characterized by calibrated formula feeding recommendations or a control group with ad lib feeds as per usual care. Intervention group parents will also be given written instructions on infant hunger and satiety cues as well as copies of videos with guidance on bottle feeding and how to soothe fussy infants without feeding. The investigators hypothesize that the calibrated formula intake intervention will reduce rapid infant gain and overweight during infancy resulting in lower weight-for-length at age 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Term or Early Term (≥37 weeks), singleton infants
* Infant birthweight ≥50th percentile based on the 2013 Fenton Growth Charts (which account for sex of child and gestational age at birth)
* Infant without substantial neonatal morbidity that would affect feeding or weight gain (e.g. known chromosomal abnormality, metabolic disorder, cleft lip/palate, etc.)
* Infant age ≤1 month
* Mothers with pre-pregnancy body mass index ≥25 kg/m2
* Mothers ≥18 years old
* Parental plan to exclusively feed infant 19-20 kcal/ounce formula upon delivery or by the start of the intervention period ~1 month after delivery
* Parental intention to have infant well child visits through age 6 months at a Division of Academic General Pediatrics practice site (Hope Drive, Elizabethtown, Nyes Road)
* English speaking parent

Exclusion Criteria:

* Infants who weigh less than their birthweight 21 days after delivery

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Paul, MD, MSc, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This may change in the future depending on results, although all individual participant data will be de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 29 | 31
Completed | 18 | 25
Not Completed | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 31 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 21 | 24 | 45
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Conditional Weight Gain Difference Between Study Groups
Description: Conditional weight gain is calculated as standardized residuals from the linear regression of weight for age at 6 months on weight for age at birth, with length for age at birth and 6 months and infant age at the 6-month visit entered as covariates.
  Note that there are no units for conditional weight gain. The CWG score represents the variation in child weight gain not explained by child age, birth length, or birth weight. A CWG score of zero represents the population mean. Positive CWG scores (above the estimated regression) indicate more rapid or faster than average weight gain, while negative scores (below the estimated regression) indicate slower weight gain. There are no maximum values.
Time Frame: Between birth and 6 months
Measure: Mean (95% Confidence Interval); unit: Conditional Weight Gain score
Groups:
- Intervention: For those with weight-for-length <75th percentile, research staff provided parents with a recommendation for total daily formula volume to be consumed based upon energy requirement (kcal/kg/day) research conducted by Butte et al. that accounts for sex, weight, and current age. To provide guidance for what parents should expect over the next month, the child's weight-for-length percentile was reviewed. Parents were informed of the volume to expect at the subsequent visit in month with the expectation that the child would maintain the same weight-for-age percentile. For those with weight-for-length ≥75th percentile, recommended current daily formula volumes were calculated based upon the child's current age, weight, and energy requirement (kcal/kg/day) with a 10% reduction in recommended daily volume. Parents were also informed of the volume to expect at the subsequent visit in one month should the child maintain the same weight-for-age percentile, again with a 10% reduction.
- Control: Usual care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 31
Conditional Weight Gain score | 0.27 [-0.20 to 0.75] | -0.12 [-0.62 to 0.37]

2. Secondary Outcome: Conditional Weight Gain Difference Between Study Groups
Description: Conditional weight gain is calculated as standardized residuals from the linear regression of weight for age at 6 months on weight for age at 1 month, with length for age at 1 month and 6 months and infant age at the 6-month visit entered as covariates.
  Note that there are no units for conditional weight gain. The CWG score represents the variation in child weight gain not explained by child age, birth length, or birth weight. A CWG score of zero represents the population mean. Positive CWG scores (above the estimated regression) indicate more rapid or faster than average weight gain, while negative scores (below the estimated regression) indicate slower weight gain. There are no maximum values.
Time Frame: During the intervention period spanning Ages 1-6 Months
Measure: Mean (95% Confidence Interval); unit: Conditional weight gain score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 30
Conditional weight gain score | 0.28 [-0.20 to 0.77] | -0.14 [-0.63 to 0.35]

3. Secondary Outcome: Mean Weight-for-Length Z-score (WLZ) on World Health Organization Child Growth Standards
Description: Weight-for-Length Z-score is based on values from the World Health Organization Growth Standards. A z-score of 0 represents the population mean. Positive values represent values above the population mean. Negative values represent values below the population mean
Time Frame: 1 time point at age 6 Months
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 25
Z-score | 0.73 [0.16 to 1.30] | 0.65 [0.28 to 1.03]

4. Secondary Outcome: Growth Trajectory (Repeated Measures of Weight-for-length on World Health Organization Child Growth Standards) During the Intervention Period
Description: repeated measures analysis of weight-for-length
Time Frame: Spanning ages 1-6 months
Measure: Mean (95% Confidence Interval); unit: kg/m
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 30
kg/m | 12.4 [12.1 to 12.7] | 12.1 [11.8 to 12.3]

5. Secondary Outcome: Percentage of Infants With Overweight (Weight-for-Length ≥95th Percentile on World Health Organization Child Growth Standards)
Description: % overweight by study group
Time Frame: 1 time point at age 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 25
Participants | 4 [6.4 to 47.6] | 2 [1.0 to 26.0]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Growth faltering defined as either:
  1. Weight-for-length <5th percentile for sex and age on the WHO growth chart
  2. Downward crossing of >2 major centile lines on the WHO growth chart (relevant major lines include 95th, 90th, 75th, 50th, 25th, 10th, 5th) after enrollment
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 12/29 | 13/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=29) | Control (N=31)
Growth Faltering (Metabolism and nutrition disorders) | 12 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT05104073/Prot_SAP_ICF_000.pdf